CLINICAL TRIAL: NCT01540357
Title: Mindfulness-based Therapy For the Treatment of Chronic Tinnitus: A Randomized Controlled Pilot Study
Brief Title: Mindfulness-based Therapy in Chronic Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Principal Investigator, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBT-TIN
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Tinnitus
Keywords: mindfulness-based therapy; chronic tinnitus;

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-based therapy (Active Comparator): Treatment was performed as group therapy at two training weekends which were separated by an interval of 7 weeks (eleven hours/weekend) and in four further two-hour sessions (week 2, 9, 18 and 22).
  Interventions: Behavioral: Mindfulness-based therapy
- Treatment after waiting time (Active Comparator): Treatment was performed after completion of the active arm.
  Interventions: Behavioral: Treatment after waiting time

INTERVENTIONS:
Behavioral: Mindfulness-based therapy — Treatment was performed as group therapy at two training weekends which were separated by an interval of 7 weeks (eleven hours/weekend) and in four further two-hour sessions (week 2, 9, 18 and 22).
  Arms: Mindfulness-based therapy
Behavioral: Treatment after waiting time — Treatment was performed after completion of the active arm.
  Arms: Treatment after waiting time

SUMMARY:
In the present randomized waiting-list-controlled study the investigators examined a specific manualized mindfulness-based therapeutic approach in the treatment of chronic tinnitus.

DETAILED DESCRIPTION:
In the current randomized waiting-list-controlled pilot study, we investigate a new manualized therapeutic approach, which is based on mindfulness- and body-psychotherapy and which has been specifically developed for the treatment of tinnitus patients (Tinnitus Atemtherapie; http://www.maria-holl.de/). Essential components of the treatment program include mindfulness, meditation, selfmassage, and breathing exercises. These components are intended to help patients use their inner resources to accept responsibility for themselves, become more self-sufficient and develop symptom acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic tinnitus (duration ≥ 6 months)
* German speaking
* Subjective tinnitus

Exclusion Criteria:

* Instable medical conditions
* Objective tinnitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in tinnitus complaints as measured by the German version of the Tinnitus Questionnaire (TQ)(Baseline versus week 9) | Baseline to Week 9

SECONDARY OUTCOMES:
Change in rating scores of German versions of the Tinnitus Handicap Inventory (Hallam) (Baseline versus week 7) | Week 7
Change in rating scores of German versions of the Tinnitus Handicap Inventory (Hallam) (Baseline versus week 9) | Week 9
Change in rating scores of German versions of the Tinnitus Handicap Inventory (Hallam) (Baseline versus week 24) | Week 24
Change in rating scores of German version of the tinnitus questionnaire (Goebel/Hiller) (Baseline versus week 7) | Week 7
Change in rating scores of German version of the tinnitus questionnaire (Goebel/Hiller) (Baseline versus week 9) | Week 9
Change in rating scores of German version of the tinnitus questionnaire (Goebel/Hiller) (Baseline versus week 24) | Week 24
Change in rating scores of German version of the Beck Depression Inventory (Baseline versus week 7) | Week 7
Change in rating scores of German version of the Beck Depression Inventory (Baseline versus week 9) | Week 9
Change in rating scores of German version of the Beck Depression Inventory (Baseline versus week 24) | Week 24
Change in rating scores of German version of the tinnitus numeric rating scales (loudness, discomfort, annoyance, distractibility, unpleasantness) (Baseline versus week 7) | Week 7
Change in rating scores of German version of the tinnitus numeric rating scales (loudness, discomfort, annoyance, distractibility, unpleasantness) (Baseline versus week 9) | Week 9
Change in rating scores of German version of the tinnitus numeric rating scales (loudness, discomfort, annoyance, distractibility, unpleasantness) (Baseline versus week 24) | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, MD, Ph.D., Principal Investigator — University of Regensburg
Locations (1):
- University of Regensburg - Dep. of Psychiatry, Regensburg, Germany

REFERENCES:
- [Background] Goebel G, Hiller W. [The tinnitus questionnaire. A standard instrument for grading the degree of tinnitus. Results of a multicenter study with the tinnitus questionnaire]. HNO. 1994 Mar;42(3):166-72. German. PMID 8175381
- [Result] Kreuzer PM, Goetz M, Holl M, Schecklmann M, Landgrebe M, Staudinger S, Langguth B. Mindfulness-and body-psychotherapy-based group treatment of chronic tinnitus: a randomized controlled pilot study. BMC Complement Altern Med. 2012 Nov 28;12:235. doi: 10.1186/1472-6882-12-235. PMID 23186556